CLINICAL TRIAL: NCT04405167
Title: Phase 1 Study of Tasquinimod Alone and in Combination With Standard Therapy for Relapsed or Refractory Myeloma
Brief Title: Tasquinimod for the Treatment of Relapsed or Refractory Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual at the time when sufficient participants were already enrolled to answer the scientific question posed by the study.
Sponsor: University of Pennsylvania (Other)
Collaborators: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 842603, UPCC 45419; UPCC 45419 (Other: University of Pennsylvania)
Record Dates: First submitted 2020-03-11; First posted 2020-05-28 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — tasquinimod; ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Open label phase 1 study with pilot expansion cohorts at the maximum tolerated dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- A1: Tasquinimod single agent dose escalation (Experimental): There are up to 5 planned dose levels, with 3 de-escalation dose levels available in case dose level 1 is determined to exceed the MTD. This arm will enroll 15-30 subjects if all dose levels are explored.
  Interventions: Drug: Tasquinimod
- A2: Tasquinimod single agent expansion (Experimental): Additional subjects will enroll in arm A2 at the MTD and optimal schedule, so that 12 subjects total who are evaluable for response will have received the MTD/optimal schedule of single agent tasquinimod. Enrollment in arm A2 will not begin until enrollment in arm A1 has been completed and a single agent MTD/optimal schedule has been established.
  Interventions: Drug: Tasquinimod
- B1: Tasquinimod+IRd dose escalation (Experimental): Dose levels will be defined according to the same tasquinimod doses as in the single agent (Arm A1) dose escalation. Enrollment in arm B1 will not begin until enrollment in arm A1 has been completed and an MTD/optimal schedule has been established for single agent tasquinimod. Initial subjects in arm B1 will be enrolled at the lower of dose level 1 or one dose level below the single agent MTD . If this initial dose level is determined to exceed the combination MTD, further subjects will be enrolled at one dose level lower. Enrollment is not planned in arm B1 at doses higher than the single agent MTD. There are 9-12 planned subjects if all dose levels are explored.
  Interventions: Drug: Tasquinimod; Drug: IRd chemotherapy
- B2: Tasquinimod+IRd expansion (Experimental): Additional subjects will enroll in arm B2 at the MTD and optimal schedule, so that 12 subjects total who are both evaluable for response and previously refractory to their most recent Imid/PI combination will have received the MTD/optimal schedule of tasquinimod in combination with ixazomib, lenalidomide, and dexamethasone. To facilitate rapid enrollment and gain more experience with the combination therapy, up to 12 additional subjects with triple-class refractory myeloma (who are not previously refractory to their most recent Imid/PI combination) may be enrolled in cohort B2. Enrollment in arm B2 will not begin until enrollment in arm B1 has been completed and a combination MTD/optimal schedule has been established.
  Interventions: Drug: Tasquinimod; Drug: IRd chemotherapy

INTERVENTIONS:
Drug: Tasquinimod — Tasquinimod will be supplied as oral capsules.
Drug: IRd chemotherapy — IRd chemotherapy with ixazomib, lenalidomide, and dexamethasone
  Other Names: Ixazomib, Lenalidomide, Dexamethasone
  Arms: B1: Tasquinimod+IRd dose escalation; B2: Tasquinimod+IRd expansion

SUMMARY:
This study is the first study of tasquinimod, an inhibitor of S100A9, in patients with multiple myeloma.

DETAILED DESCRIPTION:
Tasquinimod has previously been studied as an anti-cancer agent in patients with other cancers, including a phase 3 randomized trial in patients with metastatic prostate cancer that showed an improvement in radiographic progression-free survival. The side effect profile of tasquinimod is well-characterized based on this previous experience. This trial will establish a maximum tolerated dose and optimal schedule for administration of tasquinimod in patients with multiple myeloma and then investigate the maximum tolerated dose of tasquinimod in combination with a standard myeloma regimen of ixazomib, lenalidomide, and dexamethasone (IRd). For both single agent tasquinimod and the combination of tasquinimod with IRd, exploratory expansion cohorts will be enrolled to preliminarily characterize the antimyeloma activity of each regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. 18 years of age or older
3. Multiple myeloma (MM) diagnosed according to IMWG criteria
4. Measurable disease (this is defined differently in different arms)
5. Multiple myeloma relapsed or refractory to treatment (this is defined differently in different arms)
6. Meet certain clinical laboratory criteria
7. ECOG performance status ≤2
8. Life expectancy of at least 3 months
9. For women of childbearing potential, a negative serum or urine pregnancy test prior to study treatment.
10. For women who are not postmenopausal (12 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use two methods of contraception one of which must be highly effective
11. For men: agreement to use a barrier method of contraception for 1 month before start of study treatment, during the treatment period and for 6 months after the last dose of study treatment.

Exclusion Criteria:

1. Failure to have fully recovered (i.e. ≤ Grade 1 toxicity) from the effects of prior chemotherapy (except for alopecia)
2. Active graft versus host disease
3. Treatment with any of the following:

   1. Cytotoxic chemotherapy within 3 weeks prior to the initiation of study treatment
   2. Proteasome inhibitors, Imids, or monoclonal antibodies within 2 weeks prior to the initiation of study treatment
   3. Experimental therapy within 4 weeks or 5 half-lives, whichever is shorter
   4. Systemic corticosteroids >=10 mg prednisone or equivalent within 7 days prior to the initiation of study treatment
   5. Radiotherapy within 7 days prior to initiating study treatment
   6. Plasmapheresis within 4 weeks prior to the initiation of study treatment
   7. Tasquinimod at any time
4. Known central nervous system involvement by myeloma
5. Diagnosis of smoldering multiple myeloma
6. Diagnosis of POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
7. Active plasma cell leukemia
8. Symptomatic primary (AL) amyloidosis
9. Diagnosis of myelodysplastic syndrome or myeloproliferative syndrome
10. Active other malignancy
11. Major surgery within 4 weeks prior to initiating study treatment
12. Evidence of severe or currently uncontrolled cardiovascular condition
13. Ongoing or active systemic infection that requires systemic antibiotic or parenteral anti-infective therapy
14. Active tuberculosis, active hepatitis A, B or C virus infection, or known human immunodeficiency virus (HIV) positive
15. History of pancreatitis
16. History of malabsorption or other condition that would interfere with absorption of study drugs
17. Systemic treatment within 14 days prior to the initiation of study treatment with moderate or strong inhibitor or moderate or strong inducer of cytochrome P-3A4 (CYP3A4)
18. Need for ongoing therapy drug substances of narrow therapeutic range that are metabolized mainly by CYP3A4 (alfentanil, fentanyl, quinidine, astemizole, terfenadine, sirolimus, tacrolimus, cyclosporine, cisapride, ergotamine)
19. Need for ongoing therapy with drug substances of narrow therapeutic range metabolized mainly by CYP1A2 (duloxetine, alosetron, theophylline, tizanidine, ondansetron)
20. Ongoing treatment with warfarin, unless the INR is <=3.0.
21. For subjects enrolled on the IRd combination arms, prior dose-limiting toxicity with lenalidomide or ixazomib or absolute contraindication to concomitant thrombosis prophylaxis
22. Peripheral neuropathy grade ≥2 (NCI-CTCAE)
23. Known hypersensitivity to tasquinimod or any excipients in the study treatments
24. Pregnant or nursing (lactating) women
25. Any other condition that would, in the Investigator's judgment, contraindicate subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures
26. Prior inclusion in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Optimal Dose | approximately 3 years
  Maximum tolerated dose of single agent tasquinimod (mg).

SECONDARY OUTCOMES:
Preliminary Single-Agent Toxicity Profile | approximately 3 years
  Percentage of subjects experiencing treatment-emergent grade 3/4 adverse events during therapy with single-agent tasquinimod (using the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 5)
Preliminary Combination Therapy Toxicity Profile | approximately 3 years
  Percentage of subjects experiencing treatment-emergent grade 3/4 adverse events during therapy with tasquinimod, ixazomib, lenalidomide, and dexamethasone (using the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 5)
Preliminary Single-Agent Response | approximately 3 years
  Percentage of subjects achieving a partial response or better with single-agent tasquinimod (using the response criteria of the International Myeloma Working Group)
Preliminary Assessment of Clinical Response Combination Therapy | approximately 3 years
  Percentage of subjects achieving a partial response or better with tasquinimod, ixazomib, lenalidomide, and dexamethasone (using the response criteria of the International Myeloma Working Group)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Vogl, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan R, Satilmis H, Vandewalle N, Verheye E, Vlummens P, Maes A, Muylaert C, De Bruyne E, Menu E, Evans H, Chantry A, De Beule N, Hose D, Torngren M, Eriksson H, Vanderkerken K, Maes K, Breckpot K, De Veirman K. Tasquinimod suppresses tumor cell growth and bone resorption by targeting immunosuppressive myeloid cells and inhibiting c-MYC expression in multiple myeloma. J Immunother Cancer. 2023 Jan;11(1):e005319. doi: 10.1136/jitc-2022-005319. PMID 36650020